CLINICAL TRIAL: NCT02898038
Title: Tolerance and Acceptability of AYMES PARIS
Brief Title: Acceptability and Tolerance Study of a New Oral Nutritional Supplement (ONS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Collaborators: Alison Clark Health and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AY:SC1
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Patients established on an oral nutritional supplement, being prescribed 1-2 oral nutritional supplement (ONS) providing at least 300 kcal/day will be changed onto an equivalent prescription of AYMES PARIS for a period of 9 days.
  Interventions: Dietary Supplement: AYMES PARIS

INTERVENTIONS:
Dietary Supplement: AYMES PARIS — AYMES PARIS is a powdered, high energy, oral nutritional supplement to be mixed with milk as a drink. It provides 320 kcal and 12.2 g protein per 139 ml serving. It is a Food for Special Medical Purposes (FSMP) and must, therefore, be used under medical supervision. It is not designed as a sole source of nutrition.

SUMMARY:
Tolerance and Acceptability of new oral nutritional supplement - AYMES PARIS

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of AYMES PARIS in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference,convenience etc.

To obtain data to support an ACBS submissions for AYMES PARIS (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who are able to communicate their views regarding acceptability.
* Patients established on an oral nutritional supplement, being prescribed 1-2 ONS providing approximately 300kcal/day
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Informed consent obtained.

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Patients requiring a milk-free diet
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 of protocol for full list)
* Patients with significant renal or hepatic impairment
* Patients with swallowing impairment requiring thickened fluids
* Patients with inflammatory bowel disease or previous bowel resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
GI side effects when using AYMES PARIS | 9 DAYS
  Recording of absence/presence of any nausea, vomiting, abdominal pain, bloating / flatulence, when using AYMES PARIS as assessed by presence / absence of side effect compared to baseline period

SECONDARY OUTCOMES:
Change to bodyweight of subjects when using AYMES PARIS | 9 DAYS
  Recording of bodyweight (in kg) at start of study, start of intervention and end of intervention for comparison to investigate any trend in weight change during the intervention period compared to baseline
Compliance with prescription of AYMES PARIS | 9 DAYS
  Recording of amount of AYMES PARIS consumed by subjects compared to amount prescribed. Good compliance = >80% of prescribed being consumed. Same data collected for baseline product and compared with that of AYMES PARIS
Bowel habits of subjects when using AYMES PARIS - frequency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES PARIS, as assessed by frequency of bowel movements (number of stools per day) and compared to same data recorded during baseline period
Bowel habits of subjects when using AYMES PARIS - stool consistency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES PARIS, as assessed by consistency of stools (assessed by Bristol Stool Chart) and compared to same data recorded during baseline period

IPD SHARING:
Plan to Share IPD: No